CLINICAL TRIAL: NCT06949865
Title: Clinical Research on Optimization of Acute Levodopa Challenge Test and Exploration of New Motor Paradigm Based on the Integration of Perception Technology and Artificial Intelligence
Brief Title: AI-Enhanced Optimization of Acute Levodopa Challenge Test
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Ruijin Hospital (Other); Nanjing Medical University (Other); Second Affiliated Hospital of Soochow University (Other); Beijing Hospital (Other Government); Fujian Medical University Union Hospital (Other); Guangdong Provincial People's Hospital (Other); West China Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); China-Japan Union Hospital, Jilin University (Other); Renmin Hospital of Wuhan University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Second Affiliated Hospital of Nanchang University (Other); Xijing Hospital (Other); The Affiliated Hospital of Qingdao University (Other); The Second Affiliated Hospital of Xinjiang Medical University (Unknown); Shenzhen People's Hospital (Other); Tianjin Medical University General Hospital (Other); Qilu Hospital of Shandong University (Other); The First People's Hospital of Yunnan (Other); The First Hospital of Jilin University (Other); Tianjin Huanhu Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Wannan Medical College Yijishan Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: HX-A-2024018
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Vascular Parkinsonism; Drug-induced Parkinsonism; Corticobasal Degeneration (CBD); Parkinson Disease (PD); Dementia With Lewy Body Disease; Progressive Supranuclear Palsy(PSP); Multiple System Atrophy (MSA)
MeSH Terms: conditions — Corticobasal Degeneration; Parkinson Disease; Supranuclear Palsy, Progressive; Multiple System Atrophy | interventions — Videotape Recording

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Parkinson's disease (PD) group:: Patients with confirmed Parkinson's disease diagnosed based on the 2015 International Movement Disorder Society (MDS) Parkinson's Disease Diagnostic Criteria.
  Interventions: Other: video recording
- Multiple system atrophy (MSA) group: Patients with confirmed or probable MSA diagnosed based on the diagnostic criteria for MSA published by the International Movement Disorder Society (MDS) in 2022.
  Interventions: Other: video recording
- Progressive supranuclear palsy (PSP) group: Patients with confirmed or probable PSP diagnosed based on the diagnostic criteria of the 2017 International Movement Disorder Association PSP Collaborative Group.
  Interventions: Other: video recording
- Vascular parkinsonism (VP) group: In line with the diagnostic recommendations of vascular parkinsonism in accordance with the 2004 International Association for Movement Disorders and the 2017 Chinese expert consensus.
  Interventions: Other: video recording
- Drug-induced parkinsonism (DIP) group: Parkinsonism.
  Interventions: Other: video recording
- Corticobasal degeneration (CBD) group: Diagnosis of probable or probable CBD based on the 2019 Chinese diagnostic criteria for corticobasal degeneration.
  Interventions: Other: video recording
- Dementia with Lewy Bodies (DLB) Group: Diagnosed as probable or possible DLB based on the 2017 international DLB diagnostic criteria and the 2021 Chinese DLB diagnostic criteria.
  Interventions: Other: video recording

INTERVENTIONS:
Other: video recording — The patient's motor symptoms were recorded via video for assessment purposes.

SUMMARY:
A quantitative evaluation method was developed for Parkinson's disease and other atypical parkinonism by integrating an innovative motor paradigm with perception technologies and artificial intelligence. Combined with traditional motor paradigms and the acute levodopa challenge test, this study aims to identify diagnostic cut-off values for PD and other atypical parkinonism, explore digital biomarkers for early and differential diagnosis, and establish a corresponding diagnostic model.

ELIGIBILITY:
Inclusion Criteria:

1. Parkinson's disease (PD) group: 1. Patients with confirmed Parkinson's disease diagnosed based on the 2015 International Movement Disorder Society (MDS) Parkinson's Disease Diagnostic Criteria; 2. Patients with early-stage PD meet the Hoehn-Yahr score ≤ 2.5 points, and patients with intermediate and advanced PD meet the Hoehn-Yahr score of 2.5-5 points; 3. Subjects are 50-75 years old (including boundary values), gender is not limited; 4. Agree to undergo study-related examination evaluation and sign informed consent.
2. Multiple system atrophy (MSA) group : 1. Patients with confirmed or probable MSA diagnosed based on the diagnostic criteria for MSA published by the International Movement Disorder Society (MDS) in 2022 ;2. Subjects are 50-75 years old (including boundary values), gender is not limited; 3. Agree to undergo study-related examination evaluation and sign informed consent.
3. Progressive supranuclear palsy (PSP) group: 1. Patients with confirmed or probable PSP diagnosed based on the diagnostic criteria of the 2017 International Movement Disorder Association PSP Collaborative Group; 2. Subjects are 50-75 years old (including boundary values), gender is not limited; 3. Agree to undergo study-related examination evaluation and sign informed consent.
4. Vascular parkinsonism (VP) group: 1. In line with the diagnostic recommendations of vascular parkinsonism in accordance with the 2004 International Association for Movement Disorders and the 2017 Chinese expert consensus; 2. Subjects are 50-75 years old (including boundary values), gender is not limited; 3. Agree to undergo study-related examination evaluation and sign informed consent.
5. Drug-induced parkinsonism (DIP) group: 1. Parkinsonism; 2. Drug history, the appearance of symptoms is related to specific drugs; 3. Symptoms are reversible, and the symptoms are reduced or disappeared when the corresponding drugs are reduced; 4. Rule out other causes; 5. Subjects are 50-75 years old (including boundary values), gender is not limited; 6. Agree to undergo study-related examination evaluation and sign informed consent.
6. Corticobasal degeneration (CBD) group: 1. Diagnosis of probable or probable CBD based on the 2019 Chinese diagnostic criteria for corticobasal degeneration; 2. Subjects are 50-75 years old (including boundary values), gender is not limited; 3. Agree to undergo study-related examination evaluation and sign informed consent.
7. Dementia with Lewy Bodies (DLB) Group: 1. Diagnosed as probable or possible DLB based on the 2017 international DLB diagnostic criteria and the 2021 Chinese DLB diagnostic criteria. 2. Exhibits symptoms of Parkinsonism. 3. Subjects are aged 50-75 years (inclusive), with no gender restriction. 4. Agree to undergo study-related assessments and evaluations and signs the informed consent form.

Exclusion Criteria:

1. Cognitive dysfunction, unable to complete the study (MMSE < 23)
2. Inability to tolerate levodopa shock test
3. Patients with failure of important organs (heart, lung, liver, kidney, etc.), malignant tumors, unstable conditions and other serious internal diseases
4. Those with serious behavioral problems or mental disorders
5. Inability to sign informed consent
6. Other conditions that are considered unsuitable by the investigator to participate in this study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, participants are recruited from the multicenters across China. Participants are enrolled through outpatient assessment and screening.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy | baseline
  Using quantitative assessment methods, conduct exploratory research on new methods for early diagnosis.The test correctly identified the total proportion of individuals with and without the disease.
Diagnostic Odds Ratio | baseline
  Using quantitative assessment methods, conduct exploratory research on new methods for early diagnosis.The ratio of positive likelihood ratio to negative likelihood ratio reflects the diagnostic efficiency of the test.
Specificity | baseline
  Using quantitative assessment methods, conduct exploratory research on new methods for early diagnosis.The proportion of healthy people without a certain disease correctly identified by a diagnostic test. High specificity means that the test rarely misdiagnoses healthy people as disease patients (i.e., low false positive rate).
Negative Predictive Value | baseline
  Using quantitative assessment methods, conduct exploratory research on new methods for early diagnosis.Among all individuals who tested negative, the proportion who were truly free of the disease.
Sensitivity | baseline
  Using quantitative assessment methods, conduct exploratory research on new methods for early diagnosis.The proportion of patients with a disease correctly identified by a diagnostic test. High sensitivity means that the test rarely misses cases of disease (i.e., low false negative rate).
Positive Predictive Value | baseline
  Using quantitative assessment methods, conduct exploratory research on new methods for early diagnosis.Of all the individuals who tested positive, the proportion who actually had the disease.

SECONDARY OUTCOMES:
Negative Predictive Value | baseline
  Conduct differential diagnosis between Parkinson's disease and other Parkinsonian syndromes.Among all individuals who test negative, the proportion who are truly free of the disease.
root mean square error | baseline
  Quantify the magnitude of the prediction error
Correlation Coefficient | baseline
  Strength of the linear relationship between reflection and true results
Specificity | baseline
  Conduct differential diagnosis between Parkinson's disease and other Parkinsonian syndromes.Diagnostic tests correctly identify the proportion of healthy people who do not have a disease.
Sensitivity | baseline
  Conduct differential diagnosis between Parkinson's disease and other Parkinsonian syndromes.Refers to the proportion of patients with a disease that a diagnostic test correctly identifies.
Positive Predictive Value | baseline
  Conduct differential diagnosis between Parkinson's disease and other Parkinsonian syndromes.Of all the individuals who tested positive, the proportion who actually had the disease
Coefficient of Determination | baseline
  The proportion of variation that reflects the interpretation of the results
Diagnostic Odds Ratio | baseline
  Conduct differential diagnosis between Parkinson's disease and other Parkinsonian syndromes.The ratio of positive likelihood ratio to negative likelihood ratio reflects the diagnostic efficiency of the test.
Accuracy | baseline
  Conduct differential diagnosis between Parkinson's disease and other Parkinsonian syndromes.The total proportion of individuals with and without the disease correctly identified by the test
Intraclass Correlation Coefficient | baseline
  Conduct differential diagnosis between Parkinson's disease and other Parkinsonian syndromes.Consistency and reliability of evaluation results

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Affiliated to Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will not be publicly available, but can be shared with collaborators under specific agreements.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code